CLINICAL TRIAL: NCT04403672
Title: Performance Evaluation of RealDetect™ COVID-19 RT-PCR Kit for the Detection of SARS-CoV-2 Virus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bangladesh Medical Research Council (BMRC) (Other)
Responsible Party: Sponsor
Other Study IDs: 30005052020
Record Dates: First submitted 2020-05-24; First posted 2020-05-27 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: High Sensitivity and Specificity (With 95% Confidence Interval) of RealDetect™ COVID-19 RT-PCR Kit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive: ideSHi (CRO) investigators will be blinded to the samples provided by IEDCR. That is, ideSHi investigators will not know which of the 60 samples are positive and which of the 60 samples are negative. After RT- PCR run using RealDetect RT-PCR Kit, ideSHi will send the results to the Principal investigator. The Principal investigator will also receive IEDCR results for the same samples. Finally, the PI will compare the results from ideSHi and IEDCR and determine the sensitivity, specificity, positive predictive value and negative predictive value.
  Interventions: Device: performance evaluation study of RealDetect RT-PCR Kit for COVID-19 detection
- COVID-19 Negative: ideSHi investigators will be blinded to the samples provided by IEDCR. That is, ideSHi investigators will not know which of the 60 samples are positive and which of the 60 samples are negative. After RT- PCR run using RealDetect RT-PCR Kit, ideSHi will send the results to the Principal investigator. The Principal investigator will also receive IEDCR results for the same samples. Finally, the PI will compare the results from ideSHi and IEDCR and determine the sensitivity, specificity, positive predictive value and negative predictive value.
  In addition, 60 fresh specimens which will be tested at IEDCR will also be tested at ideSHi using RealDetect on a real time basis. These samples will also be blinded by IEDCR and sent to the testing laboratory (ideSHi). Of these 60 samples, 30 will be COVID-19 positive and 30 COVID- 19 negative samples. These fresh samples will be provided to ideSHi for testing and analysis for performance evaluation of RealDetect COVID-19 RT-PCR kit.
  Interventions: Device: performance evaluation study of RealDetect RT-PCR Kit for COVID-19 detection

INTERVENTIONS:
Device: performance evaluation study of RealDetect RT-PCR Kit for COVID-19 detection — IEDCR uses many different kits for COVID-19 detection. These kits include, (1) A*Star Fortitute Kit 2 for COVID-19 detection (Singapure), (2) Sansure Biotec Limited (China), (3) ModularDx Kit (TIB Molecular Biology, Germany, and (4) DaAn Kit (China). Among these 2 kits, A*Star Fortitude Kit 2 has been known as the best kit in IEDCR depending on its performance because it rarely generates false positive or false negative results.
  A*Star Fortitude Kit 2 is used for confirmation of any discordant results for other kits in IEDCR. That is, IEDCR uses A*Star Fortitude Kit for COVID detection as the Gold Standard. In our case, this is the main reason for the selection of this kit in order to compare the performances of RealDetect™ COVID-19 RT-PCR kit.

SUMMARY:
The novel Severe acute respiratory syndrome coronavirus 2 (SARS-C0V 2) originated in Wuhan, China in December 2019. As of April 15 2020, the virus has spread across 213 countries/territories with 1,914,916 cases and 123,010 deaths and a crude case fatality ratio (CFR) of 6.4%. In Bangladesh, the situation is also grave. As of May 14, 2020, there were 18,863 cases and 283 deaths.

In order to suppress COVID-19 transmission, it is important to diagnose COVID-19 patients, which would help in the process of quarantine and isolation of the patients and also in contact tracing. COVID-19 testing can identify the SARS-CoV-2 virus and includes methods that detect the presence of virus itself such as real time reverse-transcription-polymerase chain reaction (RT-PCR), isothermal nucleic acid amplification, antigen) and those that detect antibodies produced in response to infection. Until now, RT-PCR has been known as the best approach for - detection. It would be very useful if Bangladesh had its own locally produced RT-PCR kits, provided that the kits are no less in quality than imported kits in terms of sensitivity, specificity, price etc. The present study aims to carry out the performance evaluation of RealDetect RT-PCR Kit for COVID-19 detection.

The RealDetect™ COVID-19 RT-PCR diagnostic panel is a locally produced real-time RT-PCR test intended for the qualitative detection of nucleic acid from the SARS-CoV-2 in nasopharyngeal swab specimens collected from individuals who meet SARS-CoV-2 clinical criteria. The approach is based on the RT-PCR method which uses two (Nucleocapsid 1, Nucleocapsid 2) sets of gene-specific primers and corresponding fluorescent probes to detect two specific regions within the novel coronavirus (SARS-CoV-2) nucleocapsid protein Nucleocapsid gene. This RT-PCR panel detects SARS-CoV-2 Ribonucleic acid (RNA) specifically. The approach does not generate any false positives to other coronaviruses or human microflora. The kit also contains a primer-probe set which detects human housekeeping gene, ribonuclease Protein (RNase P). That is, the Ribonuclease Protein (RNase P) serves as an internal reference control to monitor sample collection, ribonucleic acid (RNA) extraction, and amplification.

This is a case control study. The study will analyze 120 samples (60 COVID-19 positive and 60 COVID-19 negative both fresh and frozen) from Institute of Epidemiology, Disease Control and Research (IEDCR). These specimens will be blinded before handing over to Institute for Developing Science & Health Initiatives (ideSHi) for RealDetect Kit. All samples will be analyzed by Real Time PCR System. Necessary validation will also be carried out at the COVID-19 laboratory of the Dhaka Medical College Hospital and an external validation expert will be involved. The Principal Investigator (PI) will also receive the sample information regarding positive/negative status from Institute for Epidemiology, Disease Control and Research (IEDCR) and compare ideSHi and IEDCR data. Unpaired t-test, Wilcox's test, Rank test, Compare test, Mean test, Sensitivity/Specificity test, Regression analysis and Geometric mean with 95% Confidence Interval (CI) will be used to analyze the data. It needs to conduct a univariate analysis.

DETAILED DESCRIPTION:
Considering the current global pandemic, just like any other countries it is becoming very difficult for Bangladesh to fight the COVID-19 spread. An increased number of testing is needed in Bangladesh and to cope with this demand an increase in assay kits are needed urgently in the country.

Currently we are totally dependent on imported test kits. At the time when the whole world is facing a shortage of RT-PCR test kits, import from other countries seems to be very difficult. Primarily, countries manufacturing these kits are focused on meeting the demand in their own countries first and thus those countries impose a ban on exporting these kits. So, availability of the kits will become a big problem for Bangladesh to increase testing in the country.

Secondly, due to lockdown situation worldwide, transporting these kits from another country seems second big issue we are facing right now. The kits are stranded in the airports for weeks before reaching in our country. Not to mention, the quality of the test kits is being jeopardized in the whole uncertain transportation process. The RT-PCR test kits are very temperature sensitive and maintaining the cold chain is mandatory in order to perform the test properly.

Once approved, this qualitative RT-PCR based kit can be a principal tool for Bangladesh in effective diagnosis and clinical management of COVID-19 along with collective actions made by the govt. of Bangladesh. Being developed and manufactured in Bangladesh means that there will be no shortage of testing kits during this pandemic and it will also be possible to export the kit after fulfilling domestic needs. The kit will definitely be cost-effective compared to other commercially available kits & the price will be around 30% less than the commercially available kits in the country. Current purchase price of Bangladesh govt. per test of the imported COVID-19 RT-PCR test is approx. Tk. 2780/= & RealDetect™ COVID-19 RT-PCR per test cost will be approx. Tk. 1940/=

However, this type of performance evaluation study on RT-PCR method for the detection of SARS-CoV-2 virus has not yet been done in our country. This is

the rationale why we have designed this protocol for performance evaluation of RealDetect™ COVID-19 RT-PCR kit in Bangladesh for the SARS-CoV-2 virus.

Hypothesis:

RealDetect™ COVID-19 RT-PCR will be an effective diagnostic tool for the detection of SARS CoV-2 virus using nasopharyngeal swab specimens.

Methodology:

Study type & purpose:

This is a case control study. This study is expected to validate whether the locally developed RealDetect COVID-19 RT-PCR kit is suitable for the use in Bangladesh for the detection of SARS-CoV-2 in specimens collected from suspected COVID-19 patients.

Study Population and samples Testing and analysis of a total of 120 specimens will be carried out. Of the 120 samples, 60 will be stored samples (30 COVID-19 positive samples and 30 COVID-19 negative samples) from IEDCR. The positive/negative status of the samples will be blinded before sending to ideSHi. The samples have already been stored at -80 degree Celsius in the IEDCR freezer.

In addition, 60 fresh specimens which will be tested at IEDCR will also be tested at ideSHi using RealDetect on a real time basis. These samples will also be blinded by IEDCR and sent to the testing laboratory (ideSHi) as they become available. Of these 60 samples, 30 will be COVID-19 positive and 30 COVID- 19 negative samples. These fresh samples will be provided to ideSHi for testing and analysis for performance evaluation of RealDetect COVID-19 RT-PCR kit. The PI will coordinate these activities.

IEDCR will provide ideSHi with the samples needed for the performance evaluation study of RealDetect RT-PCR Kit for COVID-19 detection. It should be mentioned here that IEDCR is the government reference laboratory for COVID-19 detection in Bangladesh. There is a MOU between ideSHi and IEDCR and these two organizations have been doing collaborative work from 2014. Thus IEDCR has been involved in this study.

To avoid biasness, ideSHi (CRO) investigators will be blinded to the samples provided by IEDCR. That is, ideSHi investigators will not know which of the 60 samples are positive and which of the 60 samples are negative. After RT- PCR run using RealDetect RT-PCR Kit, ideSHi will send the results to the Principal investigator. The Principal investigator will also receive IEDCR results for the same samples. Finally, the PI will compare the results from ideSHi and IEDCR and determine the sensitivity, specificity, positive predictive value and negative predictive value.

Study Design: Case control study.

Statistical Basis of Sample Size:

Formulae:

Variable Notations:

Α (the probability of type I error) (significance level) is the probability of rejecting the true null hypothesis (0.05) Β (the probability of type II error) (1 - power of the test) is the probability of failing to reject the false null hypothesis (0.80).

PA (proportion of discordant pairs of type A), proportion of discordant pairs of type A among discordant pairs (1/4) PD (proportion of discordant pairs) among all pairs (0.11)

Npairs, required sample size pairs 2x60=120 A matched-pair design is used, with one patient in a matched pair assigned to RT-PCR positive for COVID-19 and the other one to RT-PCR negative for COVID-19. How many matched pairs need to be enrolled in the study to have a 95% chance of finding a significant difference using a two-sided test with type I error = 0.05? So, we will use a total of 120 samples; 60 COVID-19 positive samples and 60 COVID-19 negative samples.

Diagnostic Criteria for selection of COVID-19 positive and negative specimens:

IEDCR uses many different kits for COVID-19 detection. These kits include, (1) A*Star Fortitute Kit 2 for COVID-19 detection (Singapure), (2) Sansure Biotec Limited (China), (3) ModularDx Kit (TIB Molecular Biology, Germany, and (4) DaAn Kit (China). Among these 2 kits, A*Star Fortitude Kit 2 has been known as the best kit in IEDCR depending on its performance because it rarely generates false positive or false negative results.

A*Star Fortitude Kit 2 is used for confirmation of any discordant results for other kits in IEDCR. That is, IEDCR uses A*Star Fortitude Kit for COVID detection as the Gold Standard. In our case, this is the main reason for the selection of this kit in order to compare the performances of RealDetect™ COVID-19 RT-PCR kit.

Consents from the patients are not required. Specimens will be obtained from IEDCR and so there is no requirement of patient's enrollment and consents from the patients.

All specimens will be diagnosed as COVID-19 positive on the basis RT-PCR positive results with Ct value ≤ 30 for the viral RNA. If the respiratory

specimens give positive results upon RT-PCR analysis at the lab targeting the conserved viral gene(s) for SARS-CoV-2, it will be considered as confirmed positive case for COVID-19.

On the other hand, if the respiratory specimens give negative results with no amplification upon RT-PCR analysis at the lab targeting the conserved viral gene(s) for SARS-CoV-2, it will be considered as confirmed negative case for COVID-19.

Place of study: Institute for Developing Science & Health Initiatives (ideSHi) ; Mohakhali, Dhaka.

Sample Collection Site(s): Virology Laboratory, Institute of Epidemiology, Disease Control and Research (IEDCR), Mohakhali, Dhaka

Note: IEDCR will provide ideSHi with the samples needed for the performance evaluation study of RealDetect RT-PCR Kit for COVID-19 detection. It should be mentioned here that IEDCR is the government reference laboratory for COVID-19 detection in Bangladesh. IEDCR has its own stored samples in - 80°C. There is a MOU between ideSHi and IEDCR and these two organizations have been doing collaborative work from 2014.

Data Collection Procedure: COVID-19 positive samples will be confirmed by laboratory findings of positive RT-PCR results for the viral RNA. Selection of the specimens will be carried out following the inclusion and exclusion criteria. After data collection, data will be stored in an Excel sheet for later analysis.

Data Analysis:

The sensitivity, specificity, positive predictive value and negative predictive value of RealDetect™ RT-PCR kit will be determined. Alongside sensitivity, specificity, positive predictive value and negative predictive value, Kappa coefficient, positive likelihood ratio, and negative likelihood ratio will also be calculated

Unpaired t-test, Wilcox's test, Rank test, compare test, Mean test, Sensitivity/Specificity test, Regression analysis and Geometric mean with 95% CI will be used to analyze the data. It will need to conduct a univariate analysis. A p value of ≤0.05 will be considered as the level of significant association. The sensitivity, specificity, kappa coefficient, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (LR+), negative likelihood ratio (LR-) and efficiency will be calculated using the following formulae in which TP is the number of true positives, FP the number of false positives, False negative (FN) the number of false negatives and True Negative (TN) the number of true negatives: Sensitivity = True positive (TP)/[TP + FN]; Specificity = TN/ [TN + False positive (FP)]; Kappa coefficient K=(Observed Agreement (OA)- Agreement by Chance (AC)/ (1-AC); Accuracy = [TP + TN]/ [TP + TN +FP + FN]; Positive predictive value (PPV) = TP/[TP + FP]; Negative predictive value (NPV) = TN/[TN + FN]; LR+= sensitivity/ [100 - specificity] and LR- = [100 - sensitivity]/specificity

Utilization of Results:

1. Bangladesh Medical Research Council (BMRC) ethical clearance is needed for performance evaluation study of the RealDetect™ COVID-19 RT-PCR kit.
2. This will help for further processing of RealDetect™ COVID-19 RT-PCR kit for Director General of Drug Administration (DGDA) regulations to legally market the products in Bangladesh.

Facilities:

The Principal Investigator and other investigators of the Bangladesh University of Health Sciences (BUHS) will be coordinating the evaluation and data analysis and publication. However, the testing will be carried out in a separate organization using blinded specimens from IEDCR at the ideSHi. It is one of the Government selected organizations which has been assigned for COVID-19 testing to provide services and is also a registered Contract Research Organization (CRO). The institute has international standard Biological Safety Levels (BSL) 2 plus and BSL facilities with sophisticated equipment like real time PCR machine which is required for real time RT-PCR for COVID-19 detection.

Approval of the Head of the Department/Institute:

This collaborative study will be carried out in the following institutes:

Institute of Epidemiology, Disease Control and Research (IEDCR), Mohakhali, Dhaka (For sample collection & sample storage) And Institute for Developing Science & Health Initiatives (ideSHi); Mohakhali, Dhaka (For sample analysis, data collection, data analysis)

Ethical Implications:

To avoid the biasness, the study will be blinded to ideSHi researchers who will be involved in the study.

Permission will be taken from Bangladesh Medical Research Council.

The privacy and confidentiality will be strictly maintained during and after data collection and data storage.

ELIGIBILITY:
Inclusion Criteria:

* Samples with positive RT-PCR results with Ct value ≤30 for the COVID-19 gene(s) at IEDCR will be selected as COVID-19 positive.
* Samples with negative RT-PCR results with no amplification for the COVID-19 gene(s) at IEDCR will be selected as COVID-19 negative.

Exclusion Criteria:

* Samples with equivocal/ambiguous RT-PCR results in terms of sigmoidal curve and Ct value will be excluded.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Testing and analysis of a total of 120 specimens will be carried out. Of the 120 samples, 60 will be stored samples (30 COVID-19 positive samples and 30 COVID-19 negative samples) from IEDCR. The positive/negative status of the samples will be blinded before sending to ideSHi. The samples have already been stored at -80 degree Celsius in the IEDCR freezer.
  In addition, 60 fresh specimens which will be tested at IEDCR will also be tested at ideSHi using RealDetect on a real time basis. These samples will also be blinded by IEDCR and sent to the testing laboratory (ideSHi) as they become available. Of these 60 samples, 30 will be COVID-19 positive and 30 COVID- 19 negative samples. These fresh samples will be provided to ideSHi for testing and analysis for performance evaluation of RealDetect COVID-19 RT-PCR kit. The PI will coordinate these activities.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-05-18 (Estimated); Primary Completion 2020-07-24 (Estimated); Study Completion 2020-07-24 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation of RealDetect™ COVID-19 RT-PCR kit | 2 months
  Determine Performance evaluation of RealDetect™ COVID-19 RT-PCR kit for the detection of SARS-CoV-2 virus using nasopharyngeal swab specimens collected in the nationwide COVID-19 screening program.
  RNA extraction from fresh Nasopharyngeal Swab sample in Viral Transport Medium(VTM) of COVID-19 patients from IEDCR (30 positive & 30 negative)
  Analysis of COVID-19 RNA samples using RT-PCR

SECONDARY OUTCOMES:
Reduce the price of RT-PCR based COVID-19 diagnostic test kits. | 1 month
  Supply locally manufacturer COVID-19 Reverse transcription polymerase chain reaction (RT-PCR) kit to govt. & private hospitals for diagnosis of COVID-19 patients.
  RNA extraction from frozen Nasopharyngeal Swab sample in Viral Transport Medium(VTM) of COVID-19 patients from IEDCR (30 positive & 30 negative)
  Analysis of COVID-19 RNA samples using Reverse transcription polymerase chain reaction (RT-PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Hassan, MBBS, PhD, Principal Investigator — Bangladesh University of Health Sciences
Locations (1):
- Institute of Epidemiology, Disease Control and Research (IEDCR), Mohakhali, Dhaka (For sample collection & sample storage), Institute for Developing Science & Health Initiatives (ideSHi); Mohakhali, Dhaka (For sample analysis, data collection, data analys, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Background] Hui DS, I Azhar E, Madani TA, Ntoumi F, Kock R, Dar O, Ippolito G, Mchugh TD, Memish ZA, Drosten C, Zumla A, Petersen E. The continuing 2019-nCoV epidemic threat of novel coronaviruses to global health - The latest 2019 novel coronavirus outbreak in Wuhan, China. Int J Infect Dis. 2020 Feb;91:264-266. doi: 10.1016/j.ijid.2020.01.009. Epub 2020 Jan 14. No abstract available. PMID 31953166
- See also: Novel Coronavirus (2019-nCoV): Situation Report — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200211-sitrep-22-ncov.pdf?sfvrsn=fb6d49b1_2.
- See also: Coronavirus disease 2019 (COVID-19) Situation Report-85 — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200415-sitrep-86-covid-19.pdf?sfvrsn=c615ea20_4.